CLINICAL TRIAL: NCT00248339
Title: An Open-label, Randomized Pilot Study to Compare the Effectiveness of Peginterferon-alfa-2b Plus Ribavirin to Peginterferon-alfa-2b Plus Epoetin-alfa and Two Doses of Ribavirin in the Treatment of Chronic Hepatitis C Virus Infection
Brief Title: Trial of Peg-interferon Plus Epoetin-alfa for Treatment of Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1988 WIRB
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Peginterferon; Ribavirin; Procrit; Epoetin-alpha
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): PEG-interferon-alpha-2b 1.5 μg/kg QW plus ribavirin ~13.3 mg/kg QD
  Interventions: Drug: Peginterferon-alpha-2b (PEG-Intron); Drug: Ribavirin
- 2 (Active Comparator): PEG-interferon-alpha-2b 1.5 μg/kg QW plus standard dose ribavirin, ~13.3 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
  Interventions: Drug: Peginterferon-alpha-2b (PEG-Intron); Drug: Ribavirin; Drug: Epoetin-alpha (Procrit)
- 3 (Active Comparator): PEG-interferon-alpha-2b 1.5 μg/kg QW plus high dose ribavirin, ~15.2 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
  Interventions: Drug: Peginterferon-alpha-2b (PEG-Intron); Drug: Ribavirin; Drug: Epoetin-alpha (Procrit)

INTERVENTIONS:
Drug: Peginterferon-alpha-2b (PEG-Intron) — PEG-interferon-alpha-2b 1.5 μg/kg QW plus ribavirin ~13.3 mg/kg QD
  PEG-interferon-alpha-2b 1.5 μg/kg QW plus standard dose ribavirin, ~13.3 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
  PEG-interferon-alpha-2b 1.5 μg/kg QW plus high dose ribavirin, ~15.2 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
Drug: Ribavirin — PEG-interferon-alpha-2b 1.5 μg/kg QW plus ribavirin ~13.3 mg/kg QD
  PEG-interferon-alpha-2b 1.5 μg/kg QW plus standard dose ribavirin, ~13.3 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
  PEG-interferon-alpha-2b 1.5 μg/kg QW plus high dose ribavirin, ~15.2 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
Drug: Epoetin-alpha (Procrit) — PEG-interferon-alpha-2b 1.5 μg/kg QW plus standard dose ribavirin, ~13.3 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
  PEG-interferon-alpha-2b 1.5 μg/kg QW plus high dose ribavirin, ~15.2 mg/kg QD, plus erythropoetin (PROCRIT®) 40,000 U/week.
  Arms: 2; 3

SUMMARY:
The purpose of this study is to determine if the use of epoetin-alpha will allow patients with chronic hepatitis C virus infection to be treated with higher doses of peginterferon-alpha-2b and ribavirin, thus increasing chances at lower viral levels and raising sustained virologic response.

DETAILED DESCRIPTION:
Chronic infection with hepatitis C virus (HCV) leads to cirrhosis, hepatocellular carcinoma and liver failure. The treatment for end stage liver disease is hepatic transplantation. It is therefore important the patients with chronic HCV infection be recognized and treated before they develop advanced disease. The most effective therapy for patients with chronic HCV appears to be the combination of peginterferon-alpha-2b (PEG-Intron) plus ribavirin. Overall, 54% of patients treated with these medications achieve sustained virologic response. Response to therapy is greatly enhanced in those patients who can tolerate this therapy and remain on treatment without the need for dose reduction. The single most common reason for reducing the dose of ribavirin is anemia. Ribavirin causes a dose dependent hemolytic anemia and this side effect is believed to be exacerbated by the marrow suppressive effects of interferon. Preliminary studies have suggested that anemia can be overcome with the use of erythropoetin. The present pilot study will test the hypothesis that treatment with Epoetin-alph will allow patients with chronic HCV to utilize higher doses of ribavirin along with PEG-Intron therapy and that this will lead to a more rapid decline in HCV RNA titer and an increase in sustained virologic response.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positive in serum
* HCV genotype 1
* Liver histology consistent with chronic HCV performed within 24 months prior to starting medication in this study

Exclusion Criteria:

* Previous interferon treatment
* Any other cause for liver disease
* Hemoglobin >10 gm/dl
* WBC >3,000/cubic mm
* Platelet count > 80,000/cubic mm
* Serum albumin < 3.5 gm.dl
* Conjugated serum bilirubin > 2.0 mg/dl
* INR > 1.5
* Positive HIV test
* Refusal to use adequate contraception in female subjects or the spouse.sexual partners of male subjects
* An elevation in TSH (thyroid stimulating hormone). Patients with a pre-existing thyroid disorder may enter the study if their TSH level can be maintained within the normal range.
* Women who are pregnant or breast feeding.
* A history of decompensated liver disease defined as presence of ascites, bleeding esophageal or gastric varices or hepatic encephalopathy.
* Patients with active alcohol/drug use.
* Patients with active psychiatric disorders which might be exacerbated by interferon therapy including schizophrenia and severe depression.
* Use of any immune suppressive medications within 3 months of starting interferon therapy.
* A history of cardiac disease to include recent myocardial infarction or angina.
* Patients with previous exposure to Procrit, Aranesp, GA_EPO, or any other Epoetin formulations, within 6 months prior to enrollment in this study.
* Patients with known sensitivity to mammalian cell-derived products.
* Patients with known hypersensitivity to human albumin.
* Patients unable to provide informed consent.
* Any other medical condition which the primary investigator feels might be exacerbated or jeopardise the patient's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The mean dose of ribavirin utilized in each of the 3 treatment arms will be compared. | 18 months

SECONDARY OUTCOMES:
Number of patients in each group who required a dose reduction of ribavirin | 18 months
Rate of virologic response and sustained virologic response observed in each group | 18 months
Rate of decline in HCV RNA titer in each group | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L. Shiffman, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] McHutchison JG, Gordon SC, Schiff ER, Shiffman ML, Lee WM, Rustgi VK, Goodman ZD, Ling MH, Cort S, Albrecht JK. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. N Engl J Med. 1998 Nov 19;339(21):1485-92. doi: 10.1056/NEJM199811193392101. PMID 9819446
- [Background] Poynard T, Marcellin P, Lee SS, Niederau C, Minuk GS, Ideo G, Bain V, Heathcote J, Zeuzem S, Trepo C, Albrecht J. Randomised trial of interferon alpha2b plus ribavirin for 48 weeks or for 24 weeks versus interferon alpha2b plus placebo for 48 weeks for treatment of chronic infection with hepatitis C virus. International Hepatitis Interventional Therapy Group (IHIT). Lancet. 1998 Oct 31;352(9138):1426-32. doi: 10.1016/s0140-6736(98)07124-4. PMID 9807989
- [Background] Lindsay KL, Trepo C, Heintges T, Shiffman ML, Gordon SC, Hoefs JC, Schiff ER, Goodman ZD, Laughlin M, Yao R, Albrecht JK; Hepatitis Interventional Therapy Group. A randomized, double-blind trial comparing pegylated interferon alfa-2b to interferon alfa-2b as initial treatment for chronic hepatitis C. Hepatology. 2001 Aug;34(2):395-403. doi: 10.1053/jhep.2001.26371. PMID 11481625
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Shiffman ML, Hofmann CM, Sterling RK, Luketic VA, Contos MJ, Sanyal AJ. A randomized, controlled trial to determine whether continued ribavirin monotherapy in hepatitis C virus-infected patients who responded to interferon-ribavirin combination therapy will enhance sustained virologic response. J Infect Dis. 2001 Aug 15;184(4):405-9. doi: 10.1086/322778. Epub 2001 Jul 16. PMID 11471097
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553